CLINICAL TRIAL: NCT03532646
Title: Endoscopic Complications After Roux-en Y Gastric Bypass Versus Mini/One Anastomosis Gastric Bypass
Brief Title: Endoscopic Complications After Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana Klinikum Offenbach (Other)
Responsible Party: Principal Investigator, Christine Stier, Dr. med. Sonja Chiappetta, MD, senior consultant, principal investigator, Sana Klinikum Offenbach
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FF 111/2016
Record Dates: First submitted 2018-04-24; First posted 2018-05-22 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastroscopy

STUDY DESIGN:
Intervention Model Description: All patients who underwent RYGB and MGB/OAGB readmitted for complications in our centre of excellence are getting observed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: RYGB (Other): All patients who underwent RYGB and were readmitted to upper endoscopy are getting observed
  Interventions: Procedure: upper endoscopy
- group 2:MGB/OAGB (Other): All patients who underwent MGB/OAGB and were readmitted to upper endoscopy are getting observed
  Interventions: Procedure: upper endoscopy

INTERVENTIONS:
Procedure: upper endoscopy — endoscopy of the gastrointestinal tract

SUMMARY:
Endoscopic complications such as gastro-esophageal reflux disease, ulcera, gastritis, bile reflux, anastomotic stricture and so on are described after gastric bypass surgery. The incidence of these complications after RYGB versus MGB/OAGB are getting observed.

DETAILED DESCRIPTION:
All patients who were readmitted to our centre of excellence for obesity and metabolic surgery (October 2014 - March 2018) are observed regarding endoscopic complications in s.a. RYGB and MGB/OAGB.

ELIGIBILITY:
Inclusion Criteria:

* all patients who underwent RYGB or MGB/OAGB as a primary surgery and were readmitted to tho hospital undergoing upper endoscopy are included

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Complication | Up to 15 years post surgery
  Pathological finding during upper endoscopy

SECONDARY OUTCOMES:
Weight Loss since Surgery | Up to 15 years post surgery
  Weight Loss since Surgery: Total Weight Loss in %
toxic status | Up to 15 years post surgery
  toxic status (NSAID)
toxic status II | Up to 15 years post surgery
  toxic status (nicotin)
Revisional Surgery | Up to 15 years post surgery
  Revisional Surgery due to complication

CONTACTS AND LOCATIONS:
Overall Officials: Christine Stier, MD, Principal Investigator — Sana Klinikum Offenbach/Sana Klinikum Remscheid
Locations (1):
- Sana obesity center, Remscheid, Germany

IPD SHARING:
Plan to Share IPD: No
Data will be published anonymous in a peer review journal

REFERENCES:
- [Result] De Palma GD, Forestieri P. Role of endoscopy in the bariatric surgery of patients. World J Gastroenterol. 2014 Jun 28;20(24):7777-84. doi: 10.3748/wjg.v20.i24.7777. PMID 24976715
- [Result] Abd Ellatif ME, Alfalah H, Asker WA, El Nakeeb AE, Magdy A, Thabet W, Ghaith MA, Abdallah E, Shahin R, Shoma A, Dawoud IE, Abbas A, Salama AF, Ali Gamal M. Place of upper endoscopy before and after bariatric surgery: A multicenter experience with 3219 patients. World J Gastrointest Endosc. 2016 May 25;8(10):409-17. doi: 10.4253/wjge.v8.i10.409. PMID 27247708